CLINICAL TRIAL: NCT01430104
Title: A Study to Assess the Effects on Serum Calcium When Teriparatide is Used With Active Vitamin D in Osteoporosis Patients
Brief Title: A Study of Teriparatide in Japanese Osteoporosis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14454; B3D-JE-GHDT (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-09-06; First posted 2011-09-07 (Estimated); Results first posted 2012-12-28 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2012-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teriparatide + Aspara-CA + Alfarol (Experimental): Aspara-CA 600 milligrams (mg) and Alfarol 1.0 microgram (µg) administered orally once daily throughout the study. Teriparatide 20 µg administered subcutaneously once daily for 28 days during the Treatment Period.
  Interventions: Drug: Teriparatide; Drug: Aspara-CA 600 mg; Drug: Alfarol 1.0 µg

INTERVENTIONS:
Drug: Teriparatide — Administered subcutaneously during the Treatment Period
  Other Names: LY333334; Forteo; Forsteo
Drug: Aspara-CA 600 mg — Administered orally throughout the study
Drug: Alfarol 1.0 µg — Administered orally throughout the study

SUMMARY:
The purpose of this trial is to assess the effects on serum calcium when teriparatide is used with active vitamin D in osteoporosis patients.

This study consists of a Screening Period, a 14-day Lead-in Period, a 28-day Treatment Period, and a 7-day Follow-up Period. Patients will take vitamin D and calcium supplementation from the Lead-in Period throughout the study. During the Treatment Period, daily administration of teriparatide will be added.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory Japanese males or postmenopausal females with osteoporosis, as determined by the Japanese Society for Bone and Mineral Research (JSBMR) diagnostic criteria

Exclusion Criteria:

* Prior treatment with parathyroid hormone (PTH) or any PTH analog
* History of metabolic bone disorders other than primary osteoporosis
* Fractures caused by diseases other than osteoporosis
* Abnormal thyroid function
* Hyperparathyroidism or hypoparathyroidism
* Severe or chronically disabling conditions other than osteoporosis
* Currently has or has a history of spruce, inflammatory bowel disease, or malabsorption syndrome
* Currently has, or a has a history of, nephrolithiasis or urolithiasis in the 2 years prior to screening
* Clinically significant abnormal laboratory values or electrocardiogram
* Treatment with oral bisphosphonates at any time in the 3 months prior to enrollment, treatment with any bisphosphonate for more than 60 days in the 6 months prior to enrollment, or with intravenous bisphosphonates at any time in the 24 months prior to enrollment; or in case of oral bisphosphonates administered once a week, the equivalent as the above
* Treatment with injectable calcitonin in the 3 months prior to enrollment
* Treatment with raloxifene hydrochloride for more than 3 months in the 6 months prior to enrollment
* Treatment with systemic corticosteroids, except for orally inhaled or nasally inhaled corticosteroids, in doses <= 800 micrograms per day (µg/day) beclomethasone dipropionate or equivalent in the 3 months prior to screening, or for more than 30 days in the 12 months prior to enrollment
* Treatment with anticonvulsants, except for benzodiazepines, in the 6 months prior to enrollment
* Prior treatment with strontiumranate or denosumab (anti-RANKL antibody)
* Prior external beam radiation therapy involving the skeleton
* Current or a history of malignant neoplasm in the 5 years prior to screening, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that had been definitively treated

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide: Aspara-CA (600 milligrams [mg]) and Alfarol (1.0 microgram [µg]) were administered orally once daily after the planned Teriparatide dose during the 14-day Lead-in Period and after the Teriparatide dose during the 28-day Treatment Period. Teriparatide (20 µg) was administered subcutaneously once daily for the 28-day Treatment Period.
Period: 14-Day Lead-In Period
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Started | 30
Completed | 30
Not Completed | 0
Period: 28-Day Teriparatide Treatment Period
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Started | 29 (1 participant withdrew from the study after completing the 14-day Lead-in Period.)
Received at Least 1 Dose of Teriparatide | 29
Completed | 28
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Number analyzed (Participants) | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 70 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 29
Number of Participants with Urine Calcium Excreted Over 0.3 Grams per Day (g/day) [Number; unit: participants] — Baseline calcium measures were assessed over a 24-hour period on the last day of the 14-day Lead-in Period (Day -1), after participants had been receiving Aspara-CA and Alfarol supplements, to determine the total urine calcium excreted per day.
  participants
    Urine calcium excreted >0.3 g/day | 0
    Urine calcium excreted ≤0.3 g/day | 29
Mean Urine Calcium Excreted [Mean (Standard Deviation); unit: grams per day (g/day)] — Baseline calcium measures were assessed on the last day of the 14-day Lead-in Period (Day -1), after participants had been receiving Aspara-CA and Alfarol supplements. One participant was excluded from the analysis because the participant accidentally dropped the urine collection sample during baseline (N=28).
  grams per day (g/day) | 0.12 (0.05)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serum Calcium Level Over 11.0 Milligrams Per Deciliter (mg/dL)
Description: Total serum calcium concentration adjusted by serum albumin concentration. Corrected calcium (mg/dL) = total serum calcium concentration (mg/dL) + 4.0 - serum albumin concentration (grams per deciliter [g/dL]). Postdose refers to after Teriparatide dose.
Time Frame: Day 28 (16 and 24 hours postdose)
Population: All enrolled participants who received at least 1 dose of Teriparatide and had either a 16-hour or 24-hour postdose serum calcium assessment on Day 28 were included in the analysis.
Measure: Number; unit: participants
Groups:
- 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide: Aspara-CA (600 milligrams [mg]) and Alfarol (1.0 microgram [µg]) were administered orally once daily after the Teriparatide dose during the 28-day Treatment Period. Teriparatide (20 µg) was administered subcutaneously once daily for the 28-day Treatment Period.
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Number analyzed (Participants) | 28
participants
  16 hours postdose | 0 (0)
  24 hours postdose | 0

2. Secondary Outcome: Number of Participants With Serum Calcium Level Over 11.0 Milligrams Per Deciliter (mg/dL) and 13.5 mg/dL, Respectively at Any Time Postbaseline
Description: Total serum calcium concentration adjusted by serum albumin concentration. Corrected calcium (mg/dL) = total serum calcium concentration (mg/dL) + 4.0 - serum albumin concentration (grams per deciliter [g/dL]). Serum calcium levels presented are for any time postdose on any day during the 28-day Teriparatide Treatment Period.
Time Frame: Day 1 up to Day 28 (Teriparatide Treatment Period)
Population: All enrolled participants who received at least 1 dose of Teriparatide and had at least 1 postdose serum calcium assessment were included in the analysis.
Measure: Number; unit: participants
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Number analyzed (Participants) | 29
participants
  Serum Calcium > 11.0 mg/dL | 0
  Serum Calcium > 13.5 mg/dL | 0

3. Secondary Outcome: Mean Serum Calcium Levels
Description: Daily profiles of corrected mean serum calcium levels were determined for each participant. Corrected calcium (milligram per deciliter [mg/dL]) = total serum calcium concentration (mg/dL) + 4.0 - serum albumin concentration (grams per deciliter [g/dL]). The Least Squares (LS) means were adjusted for Day, Timepoint, Day*Timepoint, and random error. At baseline, participants received only Aspara-CA and Alfarol supplements and the timepoints were based on the times before Aspara-CA and Alfarol administration (predose) and after Aspara-CA and Alfarol administration (postdose). During the 28-day Teriparatide Treatment Period, timepoints were based on before Teriparatide administration (predose) and after Teriparatide administration (postdose).
Time Frame: Baseline (Day -1 of 14-day Lead-in Period) and Day 1 and Day 7 and Day 14 and Day 28 at 0 hours (h), 2 h, 4 h, 6 h, 16 h, and 24 h postdose (28-day Teriparatide Treatment Period)
Population: All enrolled participants who received at least 1 dose of Teriparatide, completed all protocol requirements, and had at least 1 postdose serum calcium assessment were included in the analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Number analyzed (Participants) | 29
mg/dL
  Baseline: 0 h predose | 9.00 [8.92 to 9.07]
  Baseline: 2 h postdose | 9.11 [9.03 to 9.19]
  Baseline: 4 h postdose | 8.98 [8.91 to 9.05]
  Baseline: 6 h postdose | 8.92 [8.86 to 8.98]
  Baseline: 16 h postdose | 8.97 [8.90 to 9.03]
  Baseline: 24 h postdose | 8.74 [8.67 to 8.81]
  Day 1: 0 h predose | 8.74 [8.67 to 8.81]
  Day 1: 2 h postdose | 9.17 [9.10 to 9.24]
  Day 1: 4 h postdose | 9.16 [9.09 to 9.24]
  Day 1: 6 h postdose | 9.14 [9.07 to 9.21]
  Day 1: 16 h postdose | 8.85 [8.79 to 8.91]
  Day 1: 24 h postdose | 8.70 [8.64 to 8.77]
  Day 7: 0 h predose (n=28) | 9.02 [8.95 to 9.09]
  Day 7: 2 h postdose (n=28) | 9.41 [9.33 to 9.48]
  Day 7: 4 h postdose (n=28) | 9.43 [9.35 to 9.51]
  Day 7: 6 h postdose (n=28) | 9.36 [9.29 to 9.42]
  Day 7: 16 h postdose (n=28) | 9.02 [8.96 to 9.09]
  Day 7: 24 h postdose (n=28) | 8.82 [8.75 to 8.89]
  Day 14: 0 h predose (n=28) | 8.99 [8.91 to 9.06]
  Day 14: 2 h postdose (n=28) | 9.35 [9.28 to 9.43]
  Day 14: 4 h postdose (n=28) | 9.39 [9.31 to 9.46]
  Day 14: 6 h postdose (n=28) | 9.29 [9.22 to 9.36]
  Day 14: 16 h postdose (n=28) | 9.03 [8.96 to 9.09]
  Day 14: 24 h postdose (n=28) | 8.89 [8.82 to 8.96]
  Day 28: 0 h predose (n=28) | 8.98 [8.91 to 9.05]
  Day 28: 2 h postdose (n=28) | 9.41 [9.33 to 9.48]
  Day 28: 4 h postdose (n=28) | 9.42 [9.34 to 9.50]
  Day 28: 6 h postdose (n=28) | 9.33 [9.26 to 9.39]
  Day 28: 16 h postdose (n=28) | 9.04 [8.98 to 9.11]
  Day 28: 24 h postdose (n=28) | 8.85 [8.78 to 8.92]

4. Secondary Outcome: Change From Baseline in Serum Calcium
Description: Corrected calcium (milligram per deciliter [mg/dL]) = total serum calcium concentration (mg/dL) + 4.0 - serum albumin concentration (grams per deciliter [g/dL]). The Least Squares (LS) means were controlled for Day, Timepoint, Day*Timepoint, and random error. Postdose refers to after Teriparatide dose.
Time Frame: Baseline (Day -1 of the 14-day Lead-in Period), Day 1, Day 7, Day 14, Day 28 at 0 hours (h), 2 h, 4 h, 6 h, 16 h, and 24 h postdose (28-day Teriparatide Treatment Period)
Population: All enrolled participants who complied received at least 1 dose of Teriparatide, completed all protocol requirements, and had at least 1 postdose serum calcium assessment were included in the analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Groups:
- 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide: Aspara-CA (600 milligrams [mg]) and Alfarol (1.0 microgram [µg]) were administered orally once daily after the Teriparatide planned dose during 14-day Lead-in Period and after the Teriparatide dose during the 28-day Treatment Period. Teriparatide (20 µg) was administered subcutaneously once daily for the 28-day Treatment Period.
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Number analyzed (Participants) | 29
mg/dL
  Change from Baseline Day 1: 0 h predose | -0.255 [-0.317 to -0.194]
  Change from Baseline at Day 1: 2 h postdose | 0.059 [-0.006 to 0.123]
  Change from Baseline at Day 1: 4 h postdose | 0.183 [0.113 to 0.252]
  Change from Baseline at Day 1: 6 h postdose | 0.221 [0.163 to 0.278]
  Change from Baseline at Day 1: 16 h postdose | -0.117 [-0.172 to -0.062]
  Change from Baseline at Day 1: 24 h postdose | -0.038 [-0.092 to 0.016]
  Change from Baseline at Day 7: 0 h predose, n=28 | 0.018 [-0.045 to 0.080]
  Change from Baseline at Day 7: 2 h postdose, n=28 | 0.286 [0.220 to 0.351]
  Change from Baseline at Day 7: 4 h postdose, n=28 | 0.450 [0.379 to 0.521]
  Change from Baseline at Day 7: 6 h postdose, n=28 | 0.436 [0.377 to 0.494]
  Change from Baseline at Day 7: 16 h postdose, n=28 | 0.061 [0.005 to 0.117]
  Change from Baseline at Day 7: 24 h postdose, n=28 | 0.068 [0.013 to 0.123]
  Change from Baseline at Day 14: 0 h predose, n=28 | -0.018 [-0.080 to 0.045]
  Change from Baseline at Day 14: 2 h postdose, n=28 | 0.232 [0.166 to 0.298]
  Change from Baseline at Day 14: 4 h postdose, n=28 | 0.404 [0.333 to 0.474]
  Change from Baseline at Day 14: 6 h postdose, n=28 | 0.368 [0.309 to 0.426]
  Change from Baseline at Day 14: 16 h postdose,n=28 | 0.068 [0.012 to 0.124]
  Change from Baseline at Day 14: 24 h postdose,n=28 | 0.143 [0.088 to 0.198]
  Change from Baseline at Day 28: 0 h predose, n=28 | -0.021 [-0.084 to 0.041]
  Change from Baseline at Day 28: 2 h postdose, n=28 | 0.286 [0.220 to 0.351]
  Change from Baseline at Day 28: 4 h postdose, n=28 | 0.436 [0.365 to 0.506]
  Change from Baseline at Day 28: 6 h postdose, n=28 | 0.404 [0.345 to 0.462]
  Change from Baseline at Day 28: 16 h postdose,n=28 | 0.082 [0.026 to 0.138]
  Change from Baseline at Day 28: 24 h postdose,n=28 | 0.104 [0.049 to 0.159]

5. Secondary Outcome: Number of Participants With Daily Urine Calcium Excreted Over 0.3 Grams Per Day (g/Day) at Any Time Postbaseline
Description: Urine calcium levels presented are for any day during the 28-day Teriparatide Treatment Period.
Time Frame: Day 1 up to Day 28 (28-day Teriparatide Treatment Period)
Population: All enrolled participants who received at least 1 dose of Teriparatide and had at least 1 postdose urine calcium assessment were included in the analysis.
Measure: Number; unit: participants
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Number analyzed (Participants) | 29
participants | 0

6. Secondary Outcome: Mean Daily Urine Calcium Excreted
Time Frame: Day 1 and Day 7 and Day 14 and Day 28 (28-day Teriparatide Treatment Period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams per day (g/day)
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Number analyzed (Participants) | 28
grams per day (g/day)
  Day 1 | 0.13 (0.05)
  Day 7 (N=27) | 0.14 (0.05)
  Day 14 (N=27) | 0.13 (0.05)
  Day 28 (N=27) | 0.13 (0.05)

7. Secondary Outcome: Change From Baseline in Daily Urine Calcium Excreted
Time Frame: Day 1, Day 7, Day 14, Day 28 (28-day Teriparatide Treatment Period)
Population: All enrolled participants who received at least 1 dose of Teriparatide, had a baseline urine calcium assessment, and at least 1 postdose urine calcium assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: grams per day (g/day)
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Number analyzed (Participants) | 28
grams per day (g/day)
  Change from Baseline at Day 1 | 0.01 (0.02)
  Change from Baseline at Day 7 (N=27) | 0.02 (0.03)
  Change from Baseline at Day 14 (N=27) | 0.01 (0.04)
  Change from Baseline at Day 28 (N=27) | 0.01 (0.04)

8. Secondary Outcome: Concentrations of Serum 25-Hydroxy-Vitamin D
Time Frame: Day 1 (Predose, 28-day Teriparatide Treatment Period) and Day 8 and Day 15 and Day 29 (Follow-up Period) and Day 35 (Follow-up Period)
Population: All enrolled participants who received at least 1 dose of Teriparatide and had at least 1 postdose serum 25-Hydroxy-Vitamin D assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide: Aspara-CA (600 milligrams [mg]) and Alfarol (1.0 microgram [µg]) were administered orally once daily after the Teriparatide dose during the 28-day Treatment Period and after the planned Teriparatide dose during the 7-day Follow-up Period. Teriparatide (20 µg) was administered subcutaneously once daily for the 28-day Treatment Period.
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Number analyzed (Participants) | 29
nanogram per milliliter (ng/mL)
  Day 1 | 23.0 (5.4)
  Day 8 (N=28) | 22.1 (6.2)
  Day 15 (N=28) | 21.5 (6.6)
  Day 29 (N=28) | 20.1 (8.0)
  Day 35 (N=28) | 21.6 (7.2)

9. Secondary Outcome: Concentrations of Serum 1,25-Hydroxy-2-Vitamin D3
Time Frame: as for outcome 8
Population: All enrolled participants who received at least 1 dose of Teriparatide and had at least 1 postdose serum 1,25-Hydroxy-Vitamin D3 assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Number analyzed (Participants) | 29
picogram per milliliter (pg/mL)
  Day 1 | 54.0 (16.9)
  Day 8 (N=28) | 105.3 (35.2)
  Day 15 (N=28) | 108.5 (40.2)
  Day 29 (N=28) | 98.1 (32.0)
  Day 35 (N=28) | 53.9 (22.3)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected during the 28-day Teriparatide Treatment Period and the 7-day Follow-up Period.
Groups:
- 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide: Aspara-CA (600 milligrams [mg]) and Alfarol (1.0 microgram [µg]) were administered orally once daily after the Teriparatide dose during the 28-day Treatment Period and the 7-day Follow-up Period. Teriparatide (20 µg) was administered subcutaneously once daily for the 28-day Treatment Period.
Arm/Group | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 5/29
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 600 mg Aspara-CA + 1 µg Alfarol + 20 µg Teriparatide (N=29)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days